CLINICAL TRIAL: NCT00282685
Title: (Restoration of Nerve Functions by Intra-arterial Transplantation of Bone Marrow Progenitor Cells in Patients With Diabetic Poly Neuropathy (PNP)
Brief Title: Safety and Feasibility Study of Autologous Progenitor Cell Transplantation in Diabetic Neuropathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, A. M. Zeiher, Prof. Dr. med., Johann Wolfgang Goethe University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-000969-19; RENERVATE
Record Dates: First submitted 2006-01-25; First posted 2006-01-27 (Estimated); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Diabetic Neuropathies
Keywords: Patients with symmetric peripheral diabetic neuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intra-arterial stemcell therapy (Experimental): Patients were treated with intra-arterial stemcells delivered via catheter examination
  Interventions: Procedure: Intraarterial bone marrow progenitor cell transplantation

INTERVENTIONS:
Procedure: Intraarterial bone marrow progenitor cell transplantation — catheter delivery of stem cells

SUMMARY:
Treatment of patients with diabetic neuropathy by intraarterial progenitor cell transplantation.

DETAILED DESCRIPTION:
Goal is:

Stimulation of angiogenesis and induction of vasa nervorum in order to improve nerve function

ELIGIBILITY:
Inclusion Criteria:

* Patients with distal symmetrical diabetic neuropathy of the legs
* Type 1 or Type 2 Diabetes
* Stable Glucose control over last 3 months (Hba1c <7.5)
* Written informed consent

Exclusion Criteria:

* Patients with peripheral arterial disease (ABI <0.9)
* Neuropathy of other origin
* Myopathy
* Asymmetrical neuropathy
* Active infection oder fever
* Chronic inflammatory disease (z.B M. Crohn, Rheumatoid Arthritis)
* HIV or hepatitis
* Neoplastic disease without complete remission within last 5 y
* Stroke or myocardial infarction within last 3 months
* Renal failure (creatinine > 2 mg/dl)
* Liver disease (GOT > 2 upper limit or spontaneous INR > 1,5).
* Anemia (hemoglobine < 8.5 mg/dl)
* Platelets <100.000/µl
* HbA1c >7,5 %
* Allergies to Aspirin, Clopidogrel, Heparin
* Bleeding disorder
* Surgery or trauma within the last 2 months
* Pregnancy
* Mental retardation
* Participation in another study within 30 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2005-10; Primary Completion 2008-12 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Improvement of neurological score: modified NIS(LL)+7 | 1 year

SECONDARY OUTCOMES:
Modified Toronto Clinical Scoring System | 1 year
Heart rate variability | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Andreas M Zeiher, MD, Principal Investigator — Div. of Cardiology, University of Frankfurt, Germany; Dirk H Walter, MD, Study Director — Div. of Cardiology, University of Frankfurt, Germany
Locations (1):
- Div. of Cardiology and Vascular Medicine, Frankfurt, Germany